CLINICAL TRIAL: NCT05271955
Title: Medico-economic Evaluation of the Care by Serious Games in Outpatient Units and at Home for Children With Autism Spectrum Disorders
Brief Title: e-GOLIAH in Autistic Spectrum Disorders
Acronym: e-GOLIAH-ECO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP200052; 2020-A03389-30 (Other: IDRCB)
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-02

CONDITIONS: Autism Spectrum Disorder
Keywords: e-GOLIAH; e-GOLIAH-ECO; Autistic Spectrum Disorders; Children; Tablet; Games; Serious Game
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Children receiving the usual care plus intensive use of e-GOLIAH (experimental group)
  Interventions: Device: "e-GOLIAH"
- Control (Active Comparator): Children receiving only the usual treatment (control group).
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Device: "e-GOLIAH" — Usual care plus electronic tablet with games application "e-GOLIAH" (Gaming Open Library for Intervention in Autism at Home)
  Arms: Experimental
Behavioral: Usual care — Usual care which combines speech therapy, psychomotor, educational or psychological care with a developmental and / or behavioral orientation and a school life support during schooling.
  Arms: Control

SUMMARY:
Randomized open-label study comparing children aged 3 to 6 years with autism and normal cognitive development or mild cognitive impairment receiving the usual treatment plus intensive use of eGOLIAH (experimental group) with children receiving only the usual treatment (control group).

eGOLIAH (Gaming Open Library for Intervention in Autism at Home) is an accessible online platform for digital games inspired by the principles of the Early Start Denver Model (ESDM), one of the care programs validated in the management of young ASD.

The duration per patient will be one year. The exposure to e-GOLIAH for the experimental group will be done with the recommendation of intensive exposure to the game (5 sessions> ½ hour per week).

Clinical variables will be assessed at entry, 6 months and 1 year (end of study).

The EQ5D questionnaires will be collected by the supervising therapist during the follow-up visit and at the same time as the clinical variables.

DETAILED DESCRIPTION:
In a context of increasing prevalence of Autism Spectrum Disorder (ASD) and the heterogeneity of children's profiles and abilities, early diagnosis is crucial in order to implement intensive, individualized, multidimensional therapeutic care and therefore more efficient. In the context of MICHELANGELO (FP7 European Research project), we developed a serious game called GOLIAH for Gaming Open Library for Intervention for Autism at Home. Using the first beta version as functional prototype, we showed that the demonstrator could be used at home with the help of parents in addition to usual care, during a clinical study including 25 participants. Also, Billeci and colleagues showed that, after training, children's improvement in joint attention tasks was correlated with changes in brain activity and connectivity. We then developed a new version e-GOLIAH to open the opportunity to conduct a large clinical study to assess the validity of the tool in terms of children's improvements. The goals of e-GOLIAH are to bring improvements in terms of ergonomics and accessibility to this initial prototype by finalizing the tool and distributing it to therapists, parents and children with ASD, via the Curapy.com web platform. e-GOLIAH provides, in free and open access, a platform for digital games inspired by the principles of ESDM (Early Start Denver Model) allowing intensive training to improve joint attention and imitation, two key skills for early social interaction and communication. It is a more natural, child-centered intervention method practiced at home and involving parents. This innovative solution takes the assessment and management of autism care out of the usual clinical environment. eGOLIAH (Gaming Open Library for Intervention in Autism at Home) is an accessible online platform for digital games that include ten different games with different level of complexity. A key principle is the collaboration between the child and his/her parent to proceed with the games making it interactive by nature, each participant having his own tablet.

The current study e-GOLIAH-ECO is a medico-economic study powered to recruit 150 children. It is a multisite randomized open-label study comparing children aged 3 to 6 years with autism and normal cognitive development or mild cognitive impairment receiving the usual treatment plus intensive use of eGOLIAH (experimental group) with children receiving only the usual treatment (control group).

The duration per patient will be one year. The exposure to e-GOLIAH for the experimental group will be done with the recommendation of intensive exposure to the game (5 sessions> ½ hour per week).

Clinical variables will be assessed at entry, 6 months and 1 year (end of study). The EQ5D (quality of life) questionnaires will be collected by the supervising therapist during the follow-up visit and at the same time as the clinical variables.

The main objective is to evaluate the 12-month cost-effectiveness of the management of children diagnosed with ASDs using the e-GOLIAH game used at home, compared to usual management.

Secondary objective includes:

(i) To evaluate the cost-effectiveness ratio of the management of patients with ASDs using e-GOLIAH compared to usual management at 12 months of follow-up.

(ii) To explore the remaining ASD-related annual burden of the cost of disease for the two groups studied.

(iii) To evaluate the consequences of the generalization of the management of children diagnosed with ASD using e-GOLIAH, compared to a usual management, from the point of view of the Health Insurance over a period of 3 years.

(iv) To evaluate the impact of the management of children diagnosed with ASD using the e-GOLIAH game used at home, compared to usual management, on the patient's quality of life and that of their responsible parent and the correlation between the two, on adaptive symptoms, on autistic symptoms, on social interactions, on parental stress, at 6 months and at 12 months.

(v) To assess compliance with OS by children and their caregivers. The following scales will be monitored: the EQ5D-3L for quality of life, the Vineland-II scale, the Child Autism Rating Scale (CARS), the Social Responsiveness Scale (SRS), the Parenting Stress Index. In addition the medico-economic data will be monitored from regular interview and social insurance data.

ELIGIBILITY:
Inclusion criteria :

* Child with autism confirmed by a validated instrument (ADI-R or ADOS)
* Aged 3 to 6 years;
* Parent(s) agree to get involved in the constraint of using the SG 5 times / week at home for 2 periods of 3 months.
* Signature of the informed consent form by the 2 holders of parental authority or the only holder of parental authority present
* Affiliation to a social security scheme (except AME)

Non-inclusion criteria :

* Children with behavioral problems;
* Unstabilized comorbid organic pathology;
* Moderate and severe cognitive deficit (Intellectual Quotient less than 55);
* Multi or polyhandicap.
* Medication that may cause visual or cognitive impairment (PSAs, neuroleptics, etc.) or that may interfere with the study assessments
* Degenerative diseases or any other disease that could interfere with the evaluations planned during this study (known epilepsy and/or history of seizures, etc.)
* Photosensitive persons in order to avoid situations that could induce epileptic seizures in them

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of Incremental Cost-Utility Ratio (ICUR) at 12 months between the 2 groups | 12 months
  ICUR use the 5-level EQ-5D version and the child-friendly EQ-5D version (EQ5D-5L/EQ5D-Y) questionnaires (min score : 0 ; max score : 100 ; higher scores mean a better outcome)

SECONDARY OUTCOMES:
Comparison of Incremental Cost-utility ratio (ICUR) at 6 months between the 2 groups | 6 months
  ICUR use the 5-level EQ-5D version and the child-friendly EQ-5D version (EQ5D-5L/EQ5D-Y) questionnaires (min score : 0 ; max score : 100 ; higher scores mean a better outcome)
Comparison of Incremental cost-effectiveness ratio (ICER) between the 2 groups | 6 and 12 months
  ICER use the Vineland II scale (undetermined minimum and maximum)composite score, average score : 100, higher scores mean a better outcome)
Comparison of the out of pocket payment for the consumption of treatments linked to the TSA between the 2 groups | 12 months
  Amount remaining payable by the patient after deduction of reimbursements received by health insurance
Budget impact analysis (BIA) of e-GOLIAH in the management of children diagnosed with TSA for health insurance | 3 years
  Budget impact analysis (BIA) will be measured by direct resources consumed and quantified using the SNIIRAM/SNDS database
Comparison of Quality of life between the 2 groups | 6 and 12 months
  Measured by the 5-level EQ-5D version and the child-friendly EQ-5D version measured by proxy EQ-5D-5L/EQ-5D-Y(proxy) for the patient and their parent. Scale 0-100 (min score: 0, max score :100, higher scores mean a better outcome)
Comparison of Adaptive symptoms between the 2 groups | 6 and 12 months
  Use the Vineland-II Scale of socio-adaptive behavior measured by the composite score with an average to 100 of 4 dimensions: socialization, communication, life skills everyday life, and motricity (undetermined minimum and maximum composite score, average score : 100, higher scores mean a better outcome)
Comparison of Autistic symptoms between the 2 groups | 6 and 12 months
  Use the CARS (Child Autism Rating Ladder) scale, 15 items coded from 1 to 4 (score min: 0, max : 60, higher scores mean a worse outcome)
Comparison of Social interactions between the 2 groups | 6 and 12 months
  Use the SRS (Social Responsiveness Scale) scale, 65 items coded from 1 to 4 (score min: 0 ; score max : 260, higher scores mean a worse outcome)
Comparison of Parental Stress between the 2 groups | 6 and 12 months
  Use the Parental Stress Index scale, 36 items coded from 1 to 5 (score min : 0 ; max: 180, higher scores mean a worse outcome)
The child's acceptability to the e-GOLIAH game at home | 6 and 12 months
  interview with clinical team by phone contact every twice a month for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David COHEN, Professor, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (12):
- France (12):
  - Fondation Lenval - Hôpitaux Pédiatriques de Nice- CHU Lenval, Nice, Alpes Maritimes
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg, Bas-Rhin
  - Centre Hospitalier Universitaire de Toulouse, Toulouse, Haut-Garonne
  - Centre Hospitalier Universitaire de Montpellier, Montpellier, Hérault
  - Centre Hospitalier Universitaire de Tours, Tours, Indre-et-Loire
  - Centre Hospitalier Universitaire de Nancy, Nancy, Meurthe-et-Moselle
  - Centre Hospitalier d'Amiens, Amiens, Somme
  - Centre Hospitalier Universitaire de Paris - Centre Hospitalier d'Henri Laborit, Poitiers, Vienne
  - Assistance Publique - Hôpitaux de Paris, Site de la Pitié-Salpêtrière, Paris, Île-de-France Region
  - Centre Hospitalier Sainte-Anne / GHU Paris Psychiatrie et Neurosciences, Paris, Île-de-France Region
  - Assistance Publique - Hôpitaux de Paris, Site de Necker, Paris, Île-de-France Region
  - Centre Hospitalier de Versailles - André Mignot, Versailles, Île-de-France Region

REFERENCES:
- [Background] Dawson G, Rogers S, Munson J, Smith M, Winter J, Greenson J, Donaldson A, Varley J. Randomized, controlled trial of an intervention for toddlers with autism: the Early Start Denver Model. Pediatrics. 2010 Jan;125(1):e17-23. doi: 10.1542/peds.2009-0958. Epub 2009 Nov 30. PMID 19948568
- [Background] Jouen AL, Narzisi A, Xavier J, Tilmont E, Bodeau N, Bono V, Ketem-Premel N, Anzalone S, Maharatna K, Chetouani M, Muratori F, Cohen D; MICHELANGELO Study Group. GOLIAH (Gaming Open Library for Intervention in Autism at Home): a 6-month single blind matched controlled exploratory study. Child Adolesc Psychiatry Ment Health. 2017 Mar 22;11:17. doi: 10.1186/s13034-017-0154-7. eCollection 2017. PMID 28344643
- [Background] Bieleninik L, Geretsegger M, Mossler K, Assmus J, Thompson G, Gattino G, Elefant C, Gottfried T, Igliozzi R, Muratori F, Suvini F, Kim J, Crawford MJ, Odell-Miller H, Oldfield A, Casey O, Finnemann J, Carpente J, Park AL, Grossi E, Gold C; TIME-A Study Team. Effects of Improvisational Music Therapy vs Enhanced Standard Care on Symptom Severity Among Children With Autism Spectrum Disorder: The TIME-A Randomized Clinical Trial. JAMA. 2017 Aug 8;318(6):525-535. doi: 10.1001/jama.2017.9478. PMID 28787504
- [Background] Billeci L, Narzisi A, Tonacci A, Sbriscia-Fioretti B, Serasini L, Fulceri F, Apicella F, Sicca F, Calderoni S, Muratori F. An integrated EEG and eye-tracking approach for the study of responding and initiating joint attention in Autism Spectrum Disorders. Sci Rep. 2017 Oct 19;7(1):13560. doi: 10.1038/s41598-017-13053-4. PMID 29051506
- [Background] Bono V, Narzisi A, Jouen AL, Tilmont E, Hommel S, Jamal W, Xavier J, Billeci L, Maharatna K, Wald M, Chetouani M, Cohen D, Muratori F; MICHELANGELO Study Group. GOLIAH: A Gaming Platform for Home-Based Intervention in Autism - Principles and Design. Front Psychiatry. 2016 Apr 28;7:70. doi: 10.3389/fpsyt.2016.00070. eCollection 2016. PMID 27199777